CLINICAL TRIAL: NCT01589094
Title: Phase II Study of Neoadjuvant Dose Dense Gemcitabine and Cisplatin (DD GC) In Patients With Muscle-Invasive Bladder Cancer
Brief Title: Neoadjuvant Dose Dense Gemcitabine and Cisplatin (DD GC) In Patients With Muscle-Invasive Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); New York University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-071
Record Dates: First submitted 2012-04-27; First posted 2012-05-01 (Estimated); Results first posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2018-08

CONDITIONS: Bladder Cancer
Keywords: CISPLATIN; GEMCITABINE; GM-CSF; radical cystectomy; 12-071
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Gemcitabine; Cisplatin

ARMS (1):
- Gemcitabine and Cisplatin (DD GC) (Experimental): This is a Multicenter Phase II study of dose-dense (DD) gemcitabine and cisplatin (GC) neoadjuvant chemotherapy in patients with muscle-invasive bladder cancer (MIBC) who are candidates for radical cystectomy.
  Interventions: Drug: Gemcitabine and Cisplatin (DD GC)

INTERVENTIONS:
Drug: Gemcitabine and Cisplatin (DD GC) — Patients will receive six cycles of GC administered every 14 days. Gemcitabine 2,500 mg/m2 will be administered intravenously on day 1 and cisplatin 35 mg/m2 will be administered intravenously on days 1 and 2 of a 14 days cycle (with Peg GCSF). A total of six cycles of therapy will be administered followed by radical cystectomy with bilateral pelvic lymph node dissection (PLND)

SUMMARY:
The purpose of this study is to find out if standard chemotherapy (gemcitabine and cisplatin) given on a dose-dense treatment schedule (with less time between treatments) can help shrink the tumor better than standard chemotherapy given on a standard treatment schedule before the patient undergoes surgery for bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* Muscle invasive urothelial carcinoma of the bladder histologically confirmed at MSKCC or participating site ((Urothelial carcinoma invading into the prostatic stroma with no histologic muscle invasion is allowed, provided the extent of disease is confirmed via imaging and/or EUA.)
* Clinical stage T2-T4a N0/X M0 disease
* Medically appropriate candidate for radical cystectomy, as per MSKCC or participating site
* Karnofsky Performance Status ≥ 70%
* Age ≥ 18 years of age
* Required Initial Laboratory Values:
* Absolute Neutrophil Count ≥ 1000 cells/mm3
* Platelets ≥ 100,000 cells/mm3
* Hemoglobin ≥ 9.0g/dL
* Bilirubin ≤ 1.5 the upper limit of normal (ULN) for the institution
* Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN for the institution
* Alkaline phosphatase ≤ 2.5 x ULN for the institution
* Serum creatinine ≤ 1.5 mg/dL
* Estimated glomerular filtration rate ≥ 60 ml/min/1.73m2 using the CKD-EPI equation: eGFR = 141 x min(Scr/k, 1)a x max(Scr/k, 1)-1.209 x 0.993Age
* x 1.018 [if female] x 1.159 [if black] Scr is serum creatinine, k is 0.7 for females and 0.9 for males, a is -0.329 for females and -0.411 for males, min indicates the minimum of Scr/k or 1, and max indicates the maximum of Scr/k or 1
* If female of childbearing potential, pregnancy test is negative

Exclusion Criteria:

* Prior systemic chemotherapy (prior intravesical therapy is allowed)
* Prior radiation therapy to the bladder
* Evidence of NYHA functional class III or IV heart disease
* Serious intercurrent medical or psychiatric illness, including serious active infection
* Preexisting sensory grade ≥ 2 neuropathy
* Preexisting grade ≥ 2 hearing loss
* Major surgery or radiation therapy < 4 weeks of starting study treatment
* Concomitant use of any other investigational drugs
* Any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, or transient ischemic attack
* Ongoing cardiac dysrhythmias of NCI CTCAE Version 4.0 grade ≥ 2
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness or other active infection
* Concurrent treatment on another clinical trial; supportive care trials or non-treatment trials, e.g. QOL, are allowed
* Pregnancy or breast-feeding. Patients must be surgically sterile, postmenopausal, or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate. Male patients must be surgically sterile or agree to use effective contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-04; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean Bajorin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering West Harrison, Harrison, New York
  - New York University, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center@Phelps, Sleepy Hollow, New York
  - University of North Carolina, Chapel Hill, North Carolina

REFERENCES:
- [Derived] Iyer G, Balar AV, Milowsky MI, Bochner BH, Dalbagni G, Donat SM, Herr HW, Huang WC, Taneja SS, Woods M, Ostrovnaya I, Al-Ahmadie H, Arcila ME, Riches JC, Meier A, Bourque C, Shady M, Won H, Rose TL, Kim WY, Kania BE, Boyd ME, Cipolla CK, Regazzi AM, Delbeau D, McCoy AS, Vargas HA, Berger MF, Solit DB, Rosenberg JE, Bajorin DF. Multicenter Prospective Phase II Trial of Neoadjuvant Dose-Dense Gemcitabine Plus Cisplatin in Patients With Muscle-Invasive Bladder Cancer. J Clin Oncol. 2018 Jul 1;36(19):1949-1956. doi: 10.1200/JCO.2017.75.0158. Epub 2018 May 9. PMID 29742009
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine and Cisplatin (DD GC): This is a Multicenter Phase II study of dose-dense (DD) gemcitabine and cisplatin (GC) neoadjuvant chemotherapy in patients with muscle-invasive bladder cancer (MIBC) who are candidates for radical cystectomy.
  Gemcitabine and Cisplatin (DD GC): Patients will receive six cycles of GC administered every 14 days.
  Gemcitabine 2,500 mg/m2 will be administered intravenously on day 1 and cisplatin 35 mg/m2 will be administered intravenously on days 1 and 2 of a 14 days cycle (with Peg GCSF). A total of six cycles of therapy will be administered followed by radical cystectomy with bilateral pelvic lymph node dissection (PLND)
Period: Overall Study
Arm/Group | Gemcitabine and Cisplatin (DD GC)
Started | 51
Completed | 49
Not Completed | 2
Not completed — Did not receive treatment | 2

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine and Cisplatin (DD GC)
Number analyzed (Participants) | 51
Age, Continuous [Median (Full Range); unit: years] | 64 [37 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 50
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 46
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Response Rate
Description: Defined as the absence of muscle invasive carcinoma (<pT2 disease) and the absence of lymph node metastases (N0) on the final cystectomy specimen. Pathologists will assess surgical specimens systematically using criteria agreed upon for all conventional neoadjuvant treatment based on the AJCC TNM staging system.
Time Frame: 1 year
Population: 5 participants who completed 3 or more cycles of treatment did not undergo radical cystectomy: 1 refused surgery, 1 developed metastatic progression after 4 cycles, 1 withdrew consent, 1 was lost to follow-up, and 1 patient was incidentally diagnosed with moyamoya and discontinued the study because of the risk for vascular thrombotic events
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gemcitabine and Cisplatin (DD GC)
Number analyzed (Participants) | 46
percentage of participants | 57 [42 to 70]

2. Secondary Outcome: Number of Participants With Toxicity
Description: Toxicity will be graded according to the National Cancer Institute Common Toxicity Criteria for Adverse Events version 4.0.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine and Cisplatin (DD GC)
Number analyzed (Participants) | 51
Participants | 51

3. Secondary Outcome: 2 Year Recurrence Free Survival (RFS) Rate for Responders
Description: Defined as the time from treatment initiation to disease progression, local-regional or metastatic recurrence, or death analyzed using the Kaplan Meier method.
Time Frame: 2 years
Population: 26 out of 46 total participants were responders.
Measure: Number; unit: percentage of participants
Arm/Group | Gemcitabine and Cisplatin (DD GC)
Number analyzed (Participants) | 26
percentage of participants | 95

4. Secondary Outcome: 2 Year Recurrence Free Survival (RFS) Rate for Nonresponders
Description: as for outcome 3
Time Frame: 2 years
Population: 20 out of 46 total participants were responders.
Measure: Number; unit: percentage of participants
Arm/Group | Gemcitabine and Cisplatin (DD GC)
Number analyzed (Participants) | 20
percentage of participants | 52

ADVERSE EVENTS:
Time Frame: Within 30 days of study treatment, an average of 1 year
Arm/Group | Gemcitabine and Cisplatin (DD GC)
All-Cause Mortality (participants affected / at risk) | 7/51
Serious Adverse Events (participants affected / at risk) | 17/51
Other Adverse Events (participants affected / at risk) | 51/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine and Cisplatin (DD GC) (N=51)
Abdominal Pain (Gastrointestinal disorders) | 2
Creatinine Increased (Investigations) | 2
Dehydration (Metabolism and nutrition disorders) | 3
Fever (General disorders) | 1
Heart failure (Cardiac disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Infections and infestations - Other (Infections and infestations) | 2
Nausea (Gastrointestinal disorders) | 1
Pelvic infection (Infections and infestations) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1
Syncope (Nervous system disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Transient ischemic attacks (Nervous system disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Urinary tract infection (Infections and infestations) | 4
Vascular access complication (Injury, poisoning and procedural complications) | 1
Vomiting (Gastrointestinal disorders) | 3
Wound infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine and Cisplatin (DD GC) (N=51)
Anemia (Blood and lymphatic system disorders) | 44
Fatigue (General disorders) | 41
Platelet count decreased (Investigations) | 33
Alkaline phosphatase increased (Investigations) | 32
Nausea (Gastrointestinal disorders) | 32
Hyperglycemia (Metabolism and nutrition disorders) | 27
Constipation (Gastrointestinal disorders) | 22
Hypomagnesemia (Metabolism and nutrition disorders) | 21
Alopecia (Skin and subcutaneous tissue disorders) | 20
Hypocalcemia (Metabolism and nutrition disorders) | 17
Creatinine increased (Investigations) | 16
Hypoalbuminemia (Metabolism and nutrition disorders) | 15
Peripheral sensory neuropathy (Nervous system disorders) | 14
Tinnitus (Ear and labyrinth disorders) | 14
Headache (Nervous system disorders) | 12
Dysgeusia (Nervous system disorders) | 11
Urinary frequency (Renal and urinary disorders) | 11
Alanine aminotransferase increased (Investigations) | 10
Diarrhea (Gastrointestinal disorders) | 10
Mucositis oral (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 10
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Edema limbs (General disorders) | 8
Phlebitis (Vascular disorders) | 8
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8
Weight loss (Investigations) | 8
Aspartate aminotransferase increased (Investigations) | 7
Gastroesophageal reflux disease (Gastrointestinal disorders) | 7
Lymphocyte count decreased (Investigations) | 7
Cystitis noninfective (Renal and urinary disorders) | 6
Hypokalemia (Metabolism and nutrition disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Hiccups (Respiratory, thoracic and mediastinal disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 5
Anorexia (Metabolism and nutrition disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4
Blood bilirubin increased (Investigations) | 4
Blurred vision (Eye disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 4
Flatulence (Gastrointestinal disorders) | 4
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hypertension (Vascular disorders) | 4
INR increased (Investigations) | 4
Anxiety (Psychiatric disorders) | 3
Dizziness (Nervous system disorders) | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Insomnia (Psychiatric disorders) | 3
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-14): https://cdn.clinicaltrials.gov/large-docs/94/NCT01589094/Prot_SAP_000.pdf